CLINICAL TRIAL: NCT00726492
Title: A Randomised Controlled Trial Evaluating the Effects of Shortwave Diathermy and Hydrotherapy for Patients With Osteoarthritis of Their Knees
Brief Title: An Examination of the Value of Shortwave Diathermy and Hydrotherapy for Patients With Osteoarthritis of Their Knees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Dr Conor J McCarthy, Consultant Rheumatologist, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1/378/664
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2008-08-01 (Estimated); Status verified 2008-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CSWD + Hydro (Experimental): Continuous short wave diathermy and hydrotherapy
  Interventions: Other: Continuous short wave diathermy (CSWD); Other: Hydrotherapy
- Hydro alone (Experimental): Hydrotherapy alone
  Interventions: Other: Hydrotherapy
- CSWD alone (Experimental): Continuous short wave diathermy alone
  Interventions: Other: Continuous short wave diathermy (CSWD)
- Control (No Intervention): No treatment

INTERVENTIONS:
Other: Continuous short wave diathermy (CSWD) — CSWD applied twice a week for 4 weeks
  Arms: CSWD + Hydro; CSWD alone
Other: Hydrotherapy — Hydrotherapy (exercise in water) attended twice a week for 4 weeks
  Arms: CSWD + Hydro; Hydro alone

SUMMARY:
Osteoarthritis, a common disorder increasing in prevalence with advancing age, is particularly debilitating when the knees are affected. This study examined the value of hydrotherapy (exercise in water) and continuous short-wave diathermy (an electrical deep heat treatment) for the relief of osteoarthritic symptoms.

DETAILED DESCRIPTION:
Osteoarthritis is a common disabling disorder increasing in prevalence with advancing age (Blixen and Kippes, 1999). As there is a rapid increase in the percentage of people over 55 years in Western countries (Okma-Keulen and Hopman-Rock, 2001) it has become increasingly important to address issues which relate to older people. In 2010, the projected percentage of the population aged 60 years or older in Europe will be approximately 25%. The increased incidence of arthritis among older people, which is a significant health care problem today, is set to become an even greater concern in the coming years (Reginster, 2002). Rheumatic diseases are a huge encumbrance on the health care systems of countries worldwide and account for significant disability, lost productivity and reduction in quality of life (Sangha, 2000). The burden of disease relates not only to its prevalence but also to the cost of the disease to the health care system of the country, these costs include direct costs, such as the costs associated with drugs, medical care, hospitals, research, pensions and benefits and indirect costs, such as premature mortality and chronic disability (Reginster, 2002). Neither census statistics nor statistics from the Department of Health and Children revealed the true prevalence of osteoarthritis in Ireland. A search was also carried out using the Hospital Inpatient Enquiry (HIPE) system of The Economic and Social Research Institute of Ireland (ESRI) which likewise did not reveal the frequency of osteoarthritis in the population.

Osteoarthritis is characterised by progressive loss of articular cartilage, appositional subchondral bone development and osteophyte formation at the joint margins. The resulting pain, stiffness and functional limitations (Jakobsson and Hallberb, 2002) lead to diminished quality of life. The knee is a particularly common site of involvement in osteoarthritis. Osteoarthritic knee pain has been found to be associated with poor perceived health and significant disability, while psychological distress strongly associates with both pain and disability (O'Reilly et al, 1998; Sangha, 2000). Restricted knee joint mobility, in particular flexion appears to be an important determinant of disability in patients with osteoarthritis (Steultjens et al, 2000). Minor et al (1999) noted that lower extremity impairments in older adults have been linked to the reduced ability to use public transportation, climb stairs, perform household chores, shop and engage in leisure activities. Similarly van Barr (1998) noted that disability in patients with lower limb osteoarthritis is significantly related to pain and joint range of motion. Due to the chronic nature of osteoarthritis, physical modalities, lifestyle modification and patient self-management in terms of education and exercise are considered important approaches to treatment (Sangha, 2000).

Physiotherapists have an important role to play in the clinical management of osteoarthritis (Green et al, 1993) however, the effect of their involvement has rarely been assessed in terms of randomised controlled trials. Chard et al (2000) examined the research output in relation to a number of physiotherapy interventions available to patients with osteoarthritis of their knees and established that between 1950 to 1998 only 60 research articles were published, the majority of which occurred between 1985 and 1998. Advice (Maurer et al, 1999; Manek and Lane, 2000) and exercise (Puett and Griffin, 1994; Clarke, 1999; O'Reilly et al, 1999) have been clearly identified as beneficial in terms of relieving the impairments experienced by individuals with knee osteoarthritis. Indeed there is a some evidence supporting the use of a number of physiotherapy interventions including hydrotherapy (Ahern et al, 1995; Norton et al 1997; Alexander et al, 2001) and continuous short-wave diathermy (CSWD) (Wright, 1964; Lankhorst et al, 1982) for the treatment of knee osteoarthritis but there are difficulties regarding the design of many of these studies thus undermining the conclusions that have been drawn. This study presents the results of a randomised controlled factorial trial (Polger and Thomas, 2000) designed to examine hydrotherapy and/or continuous short wave diathermy (CSWD) for patients with knee osteoarthritis while also examining the perceptions of patients participating in a physiotherapy programme.

ELIGIBILITY:
Inclusion Criteria:

* Patients had to have a documented diagnosis of osteoarthritis of their knees.
* Patients had to be between 50 and 70 years inclusive.
* Patients had to have X-ray evidence of osteoarthritis of their knees.

Exclusion Criteria:

* Patients with another rheumatological condition other than osteoarthritis.
* Patients who were unable to understand the concepts, assessment and treatment involved.
* Patients who had received a cortisone injection into the knee in the previous 30 days.
* Patients for whom CSWD or hydrotherapy has been contraindicated.
* Patients who have had either CSWD or hydrotherapy in the past.
* Patients who had undergone a surgical procedure on either lower limb in the past 6 months.
* Patients who were receiving other physiotherapy treatment.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2001-06; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test | 4 and 8 weeks

SECONDARY OUTCOMES:
Visual analogue pain scale (10 cm line) | 4 and 8 weeks
Knee range of motion | 4 and 8 weeks
Arthritis Impact Measurement Scale 2 (AIMS 2) | 4 and 8 weeks
Patient interview | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tara Cusack, MMedSc PhD, Principal Investigator — University College Dublin; Conor J McCarthy, MD, Principal Investigator — Mater Misericordiae University Hospital; Leslie Daly, BSc MSc PhD, Principal Investigator — University College Dublin; Mary F McAteer, MEd PhD, Principal Investigator — University College Dublin
Locations (1):
- Mater Misericodriae University Hospital, Dublin, Dublin, Ireland